CLINICAL TRIAL: NCT05483621
Title: Hormonal Stimulation of Spermatogenesis in Non-obstructive Azoospermia
Brief Title: Hormonal Stimulation of Spermatogenesis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Abd-Elmo'men
Record Dates: First submitted 2022-07-31; First posted 2022-08-02 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Azoospermia, Nonobstructive
MeSH Terms: conditions — Azoospermia, Nonobstructive | interventions — Chorionic Gonadotropin, beta Subunit, Human

STUDY DESIGN:
Intervention Model Description: to evaluate the effect of hormonal stimulation for patients with non-obstructive azoospermia
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hormonal therapy Group (Experimental): Administration of hormonal therapy (as Beta HCG (5000 IU I.M) twice weekly for three months
  Interventions: Drug: Beta-hCG
- L-carnitine Group (Control) (Other): Administration of L-carnitine 1000 mg twice daily for three months
  Interventions: Drug: Beta-hCG

INTERVENTIONS:
Drug: Beta-hCG — Treatment of spermatogenesis

SUMMARY:
Urologists and reproductive specialists are often challenged when facing patients with severe male infertility scenarios. In particular, the treatment of men with NOA demands a deeper insight. In such cases, .

DETAILED DESCRIPTION:
The hormonal stimulation of spermatogenesis is still being explored. Thus, there is still little knowledge regarding the type of patient who might benefit from medical treatment, the optimal medication,

the regimen, and the duration of treatment. In male infertility, the induction for treatment with follicle stimulating hormone (FSH) in the induction and maintenance of spermatogenesis in patient with hypogonadotopic hypogonaism. As these patients are normally azoospermic without gonadotropin stimulation and during testosterone therapy

The presence of high numbers of progressively motile and normally formed sperms in the ejaculate during exogenous gonadotropin therapy might result in the desired clinical pregnancy for many infertile couples on an experimental basis and in some places already in clinical routine. FSH preparation are also used for treatment of normogonadotopic infertile men with idiopathic impairment of spermatogemesis.

Pulstile GnRH or exogenous gonadotropins are usually used to induce spermatogenesis and promote testicular enlargement .The regimen for gonadotropin replacement includes an initial use of human chorionic gonadotropin (HCG) for 6 to 12 months and then addition of FSH or human menopausal gonadotropins (HMG) until pregnancy

ELIGIBILITY:
Inclusion Criteria:

* Men with primary infertility due to non-obstructive azoospermia in two seminal analysis

Exclusion Criteria:

1. Patients with non-obstructive azoospermia with normal or low level of FSH.
2. Patients with serum testosterone lower than 3 nmol/L.

Ages: 19 Years to 72 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Hormonal treatment | from baseline up to 3 months after the treatment day.
  About 100 participants receiving Beta HCG (5000 IU I.M) twice weekly to evaluate the effect of hormonal stimulation for patients with non-obstructive azoospermia

CONTACTS AND LOCATIONS:
Locations (1):
- Urology department - faculty of medicine, South Valley university, Qina, Egypt

IPD SHARING:
Plan to Share IPD: Undecided